CLINICAL TRIAL: NCT00317447
Title: Oral Steroids in the Treatment of Acute Sciatica A Randomized Controlled Study
Brief Title: The Efficacy of Oral Steroids in the Treatment of Acute Sciatica
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oral Steroid Tx Acute Sciatica
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2006-04

CONDITIONS: Sciatica
Keywords: Sciatica; Lower back pain; Prednisone; Randomized, controlled clinical trial
MeSH Terms: conditions — Sciatica; Low Back Pain | interventions — Prednisone

INTERVENTIONS:
Drug: Oral Prednisone

SUMMARY:
Sciatica (lumbosacral radiculopathy) is a common diagnosis in primary care, occurring in approximately one percent of all patients with acute low back pain. (1, 2) Traditional treatment generally involves pain control (acetominophen, NSAID's, or narcotics), activity as tolerated, and time. (1, 3-8 ) The general consensus is that fifty percent of patients with sciatica recover within six weeks, and that ninety percent are better in twelve weeks.(4, 8) Those patients with intractable pain or progressive neurologic symptoms usually receive epidural steroid injections and, if necessary, decompressive laminectomy or discectomy. (2, 8, 9)

Low back pain and sciatica result in tremendous losses to our society in terms of decreased productivity and cost of treatment. (1, 12) Oral steroids are inexpensive and relatively safe medications that, if effective in reducing the pain and disability associated with sciatica, could improve the quality of patients' lives, and result in significant cost savings to society at large. We hypothesize that the use of oral steroids to treat acute sciatica will speed patients' recovery as measured by: changes in physical findings, rates of return to work and activities of daily living, pain and disability assessment scores, and decreases in the use of narcotic and non-steroidal anti-inflammatory drugs (NSAID's), and in the need for epidural injection or surgical intervention.

DETAILED DESCRIPTION:
Inclusion Criteria

To be included in this study patients had to have a diagnosis of acute sciatica as determined by the principle investigator based on the following criteria: unilateral leg pain extending below the knee (with or without strength, sensory, or reflex changes), and a positive straight leg raising sign (defined as as pain radiating from the buttock to below the knee with elevation of the leg between zero and sixty degrees). Patients had to be between twenty and sixty years of age, and had to be entered in [recruited into] the study within one week of the onset of their symptoms.

Exclusion Criteria

Patients were excluded from the study if they were pregnant or had a history of diabetes, renal failure, upper gastro-intestinal bleed, or major psychiatric disease. Patients also had to be free of symptoms suggesting more serious underlying disease as defined by the United States Agency for Healthcare Policy Research document: "Acute Low Back Problems In Adults". (11) "Red Flag" symptoms" included: a history of cancer, unexplained weight loss, fever or chills, night sweats, a history of intravenous drug use, saddle anesthesia, bowel or bladder incontinence, bone pathology, or a Neurologic emergency. Additionally, patients could be excluded for any condition that the principle investigator thought might jeopardize their safety.

Randomization and Blinding

Once the diagnosis of acute sciatica had been confirmed, subjects were randomized to receive either a nine day tapering course of prednisone or placebo capsules. The principle investigator and research nurse were blinded as to group assignment. All subjects received current standard therapy for sciatica, including: a NSAID (ibuprofen, naproxen, etodolac, or nambumetone), narcotics if needed (hydrocodone, propoxyphene, oxycodone, or morphine), activity as tolerated, and a referral for physical therapy.

Study Design

Upon entering the study all patients underwent physical exam with attention to: straight leg raising test (positive or negative), contralateral straight leg raising (positive or negative), knee and ankle stretch reflexes (0-3+), foot sensation (normal or decreased), strength (0-5) of quadriceps, foot dorsiflexors, foot plantar flexors, and ability to perform five heel lifts (0-5). Patients also completed three written instruments: a "12 Item Health Status Questionnaire" (13), a "Roland-Morris Disability Questionnaire" (14), and a "Roland-Morris Pain Rating Scale" (14). Also noted at the intake visit and each subsequent visit were the number of hours each patient was working or, if they were not employed or were retired, their estimated percent of daily living activities they were able to accomplish. Lastly, note was made of whether the patient had undergone epidural steroid injection or surgical intervention since the previous visit. Each patient underwent the same exam and completed the same questionnaires weekly for four weeks post recruitment, and then monthly for five months. This led to a total of 6 months of follow-up.

All patients received non-steroidal anti-inflammatory medication and narcotic medication if needed for pain control. Patients randomized to the study group received tapering course of prednisone: 60 mg for three days, 40 mg for three days, and 20 mg for three days. Patients randomized to the control (placebo) group received capsules identical in appearance to the prednisone capsules but containing an inert filler substance. Patients were questioned at each visit to determine whether they were taking their study medication (first nine days of the study) and whether they were still taking non-steroidal or narcotic medication (entire study).

Patients were encouraged to begin non-weight-bearing aerobic activities such as swimming and/or bike riding as soon as their pain had subsided to a reasonable degree. At this point, patients generally also referred to see a physical therapist.

Patients who had rapid improvement and were under fifty generally did not have any imaging studies performed. Project staff ordered plain films of the lumbosacral spine for most patients over age 50 . Irrespective of age, patients who had intractable pain or progressive neurologic symptoms generally had plain films of the lumbosacral spine done and also underwent magnetic resonance imaging (MRI). A separate analysis of pain level ratings, narcotic and NSAID use, and return to work rates, was performed for this subgroup with the thought that they probably represented patients with the most severe nerve root inflammation and that the effects of oral prednisone might be more or less obvious in this group.

Statistical power analysis

Statistical power analysis was performed with the primary outcome of return to work within 14 days of the intervention. The proportion of the control group returning to work was hypothesized to be 50%. Oral prednisone was hypothesized to have a 50% treatment effect, resulting in a 75% rate of return to work within 14 days. Using chi square with continuity correction, statistical power analysis found that a (study and control group) sample size of 80 per subgroup would have a power of 88% to find this difference (i.e., between 50% and 75%)statistically significant at p<.05.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of acute sciatica as determined by the principle investigator based on the following criteria:

unilateral leg pain extending below the knee (with or without strength, sensory, or reflex changes); and

a positive straight leg raising sign (defined as as pain radiating from the buttock to below the knee with elevation of the leg between zero and sixty degrees)

recruited into the study within one week of the onset of symptoms

Exclusion Criteria:

Current pregnancy

A history of:

diabetes renal failure upper gastro-intestinal bleed major psychiatric disease

Presence of any 'red flag' symptoms suggestive of more serious underlying disease as defined by the United States Agency for Healthcare Policy Research document: "Acute Low Back Problems In Adults" (11) including:

a history of cancer

unexplained weight loss

fever or chills

night sweats

a history of intravenous drug use, saddle anesthesia, bowel or bladder incontinence, bone pathology, or a Neurologic emergency.

Any condition that the principle investigator thought might jeopardize the patient's safety

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Start 2002-02; Study Completion 2004-04

PRIMARY OUTCOMES:
Physical examination findings:
straight leg raising test (positive or negative)
contralateral straight leg raising (positive or negative)
knee and ankle stretch reflexes (0-3+)
foot sensation (normal or decreased)
strength (0-5) of quadriceps
foot dorsiflexors
foot plantar flexors
ability to perform five heel lifts (0-5)
Written instruments:
HSQ 12 (Health Status Questionaire)(13)
Roland-Morris Disability Questionaire (14)
Roland-Morris Pain Rating Scale (14)

SECONDARY OUTCOMES:
Number of hours/week of work
Estimated percent of daily living activities subjects were able to accomplish
Epidural steroid injection
Surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard Holve, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser-Permanente, Santa Rosa, California, United States

REFERENCES:
- [Background] Frymoyer JW. Back pain and sciatica. N Engl J Med. 1988 Feb 4;318(5):291-300. doi: 10.1056/NEJM198802043180506. No abstract available. PMID 2961994
- [Background] Scheer SJ, Radack KL, O'Brien DR Jr. Randomized controlled trials in industrial low back pain relating to return to work. Part 2. Discogenic low back pain. Arch Phys Med Rehabil. 1996 Nov;77(11):1189-97. doi: 10.1016/s0003-9993(96)90147-1. PMID 8931535
- [Background] USDHHS, Agency for Health Care Policy and Research. Acute low back problems in adults. Rockville, MD: AHCPR; 1994. AHCPR pub number 95-0642
- [Background] Daniels JM 2nd. Treatment of occupationally acquired low back pain. Am Fam Physician. 1997 Feb 1;55(2):587-96, 601-2. PMID 9054226
- [Background] Deyo RA. Conservative therapy for low back pain. Distinguishing useful from useless therapy. JAMA. 1983 Aug 26;250(8):1057-62. PMID 6224032
- [Background] Deyo RA. Back pain revisited. Newer thinking on diagnosis and therpapy. Consultant 1993 Feb:88-97
- [Background] Griffin G, Tudiver F, Grant WD. Do NSAIDs help in acute or chronic low back pain? Am Fam Physician. 2002 Apr 1;65(7):1319-21. No abstract available. PMID 11996413
- [Background] Weber H. The natural history of disc herniation and the influence of intervention. Spine (Phila Pa 1976). 1994 Oct 1;19(19):2234-8; discussion 2233. doi: 10.1097/00007632-199410000-00022. PMID 7809761
- [Background] Kraemer J. Natural course and prognosis of intervertebral disc diseases. International Society for the Study of the Lumbar Spine Seattle, Washington, June 1994. Spine (Phila Pa 1976). 1995 Mar 15;20(6):635-9. doi: 10.1097/00007632-199503150-00001. PMID 7604337
- [Background] Guo HR, Tanaka S, Halperin WE, Cameron LL. Back pain prevalence in US industry and estimates of lost workdays. Am J Public Health. 1999 Jul;89(7):1029-35. doi: 10.2105/ajph.89.7.1029. PMID 10394311
- [Background] Radosevich DM. An abbreviated health status questionnaire: the HSQ12. The Newsletter of the Health Outcomes Institute. 1995;2:1-4
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Elashoff JD, NQuery Advisor Version 2.0, 2000, Statistical Solutions, Saugus MA